CLINICAL TRIAL: NCT05838586
Title: Sex Differences in the effecTs of brEaking uP Sedentary Behavior on vascUlar Function in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STEP Up T2D
Record Dates: First submitted 2023-04-13; First posted 2023-05-01 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants will complete three interventions in a randomized order, separated by >=6 and <90 days. The interventions are:
  1. 4 hours of prolonged SB (control, CON)
  2. 4 hours of SB broken up by 5 minutes of self-paced walking every hour (BREAK)
  3. 4 hours of SB with one 20-minute bout of self-paced walking (BOUT)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CON (Experimental): Control group
  Interventions: Behavioral: prolonged SB
- Break (Experimental)
  Interventions: Behavioral: SB broken 1
- BOUT (Experimental)
  Interventions: Behavioral: SB broken 2

INTERVENTIONS:
Behavioral: prolonged SB — 4 hours of prolonged SB
  Arms: CON
Behavioral: SB broken 1 — 4 hours of SB broken up by 5 minutes of self-paced walking every hour
  Arms: Break
Behavioral: SB broken 2 — 4 hours of SB with one 20-minute bout of self-paced walking
  Arms: BOUT

SUMMARY:
Type 2 diabetes (T2D) confers a high risk of cardiovascular disease (CVD), particularly among older adults who tend to be physically inactive. Prolonged sedentary behavior (SB) has been shown to negatively influence markers of cardiovascular risk (e.g., blood glucose, blood pressure), even among individuals who are physically active. Most studies that have examined the effects of breaking up SB have focused on young healthy males and prioritized glycemic outcomes. Additionally, sex differences in these outcomes have not been adequately examined. The present study will address these gaps. This 3-arm crossover randomized controlled trial will compare the effects of 3 SB conditions on markers of vascular function. The 3 conditions are: 1) 4 hours of prolonged SB, 2) 4 hours of SB broken up by 5 minutes of self-paced walking every hour, and 3) 4 hours of SB with one 20-minute bout of self-paced walking. In addition to examining the overall effects of each condition, sex differences in physiological responses will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* Postmenopausal (females only, ≥12 months without a menstrual period)
* Type 2 diabetes (hemoglobin A1c ≥6.5% and/or previous diagnosis of type 2 diabetes)
* ≥6 hours/day sedentary (assessed via IPAQ)
* Willingness to abstain from food, caffeine, alcohol and exercise for >= 24 hours, and tobacco/smoking for ≥12 hours prior to each intervention visit
* Ability to speak and read English

Exclusion Criteria:

* Type 1 diabetes
* Uncontrolled hypertension (resting systolic ≥160 or diastolic ≥110 mmHg)
* Initiation of hormone therapy or change in hormone therapy dose/frequency/route of administration in the previous 3 months
* Renal dialysis
* History of deep vein thrombosis (DVT)
* Evidence of cognitive impairment that could impact ability to consent and/or participation (Mini-Cog score <3)
* Achieving physical activity guidelines (≥150 minutes of MVPA/week, assessed via IPAQ))
* Physical impairment or disability that interferes with ability to engage in PA (e.g., severe osteoarthritis, lower extremity amputation [other than toe(s)/partial foot], use of a walker or wheelchair, etc.),
* Unstable medical/psychiatric condition that could impact study participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
iAUC of SBP | 90 days
  Net incremental area under the curve (iAUC) of systolic blood pressure (SBP)

SECONDARY OUTCOMES:
Net iAUC of DBP | 90 days
  Net iAUC of diastolic blood pressure
Net iAUC of of MAP | 90 days
  Net iAUC of mean arterial pressure
Net iAUC of HR | 90 days
  Net iAUC of heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Mary O Whipple, PhD, RN, PHN, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States